CLINICAL TRIAL: NCT00681018
Title: Feeding Study in Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mead Johnson Nutrition (Industry)
Responsible Party: Carol Lynn Berseth, M.D., Mead Johnson
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 3379-1
Record Dates: First submitted 2008-05-15; First posted 2008-05-20 (Estimated); Last update posted 2010-08-31 (Estimated); Status verified 2010-08

CONDITIONS: Premature Infants
Keywords: premature; infants
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Liquid human milk fortifier
  Interventions: Other: Liquid human milk fortifier
- 2 (Active Comparator): Powder human milk fortifier
  Interventions: Other: Powder human milk fortifier

INTERVENTIONS:
Other: Liquid human milk fortifier — Liquid human milk fortifier added to human milk
  Other Names: No other names -- experimental product
  Arms: 1
Other: Powder human milk fortifier — Powder human milk fortifier added to human milk
  Other Names: Enfamil Human Milk Fortifier
  Arms: 2

SUMMARY:
To evaluate weight gain of preterm infants fed fortified human milk.

ELIGIBILITY:
Inclusion Criteria:

* premature infant
* birth weight less than/equal to 1250 g
* exclusively breast fed

Exclusion Criteria:

* metabolic or chronic disease
* major surgery
* ventilator dependent

Max Age: 40 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 143 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Weight gain | 28 days

SECONDARY OUTCOMES:
Feeding tolerance | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Carol Lynn Berseth, MD, Study Director — Mead Johnson Nutrition
Locations (13):
- United States (13):
  - The University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of Florida, Jacksonville, Florida
  - Plantation General Hospital, Plantation, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Advocate Hope Children's Hospital, Oak Lawn, Illinois
  - Advocate Lutheran General Children's Hospital, Park Ridge, Illinois
  - Children's Hospital, Omaha, Nebraska
  - Queen's Hospital, Jamaica, New York
  - Pitt County Memorial Hospital, Greenville, North Carolina
  - SEAHEC, Wilmington, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Fairfax Hospital, Falls Church, Virginia
  - Virginia Commonwealth University, Richmond, Virginia